CLINICAL TRIAL: NCT04422704
Title: Mixed Study on the Impact of a Technology-based Intervention With Retired People
Brief Title: A Technology-based Intervention With Retired People
Acronym: Tech-Retired
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Nieto Riveiro (Other)
Responsible Party: Sponsor-Investigator, Laura Nieto Riveiro, Professor PhD, Universidade da Coruña
Organization: Universidade da Coruña (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/576
Record Dates: First submitted 2020-05-03; First posted 2020-06-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Aging; Retirement
Keywords: Older adults; Technological devices; Technology; Healthy Lifestyle; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retired people (Experimental): People who are either ordinarily or early retired and who have previously held a paid employment.
  Interventions: Behavioral: Technology-based-Intervention

INTERVENTIONS:
Behavioral: Technology-based-Intervention — The intervention is intended to address the concerns and needs that emerge from the participants' interviews. The intervention is based on the principles of the process of adaptation to retirement defined by Atchley and the Prochaska and Diclemente Model on the phases of preparation for retirement. The material to be used will be based on existing resources for retired people, awareness through multimedia material and knowledge of possible contributions of different technological devices to the retirement process.
  The sessions consisted of showing different exercises and devices to perform physical activities, cognitive training, relaxation activities, counselling about healthy eating and leisure-time activities.

SUMMARY:
The main objective of the study is to understand retired people's perception of retirement, to know their personal experience and to jointly seek solutions to the needs and problems encountered.

Secondarily, the aim is to understand the impact that an active aging program intervention implemented in retired people, based on the use of technology and considering the basis for the adaptation of the Prochaska and Diclemente Trans-Theoretical Model, can have in their quality of life.

DETAILED DESCRIPTION:
The present study has been approached from a mixed-methods research. Mainly, the study is focused on a Research-Action-Participation method in order for empowering and to people having more control over their lives. This approach was used taking into account the many changes caused by leaving working life to begin the stage of retirement. In reference to participatory methods, techniques such as brainstorming, and consensus-building and visual techniques have been included.

The quantitative approach is a complementary method to the qualitative approach based on a quasi-experimental study, as no control group has been introduced. From this approach, a descriptive and comparative study has been carried out on quality of life and the behavior adopted in the adaptation to retirement, both measured before and after the intervention.

The intervention program developed consists of a brief-intervention about 5 sessions lasting between 45-60 minutes. It was intended to address the concerns and needs that emerge from the participants' interviews. The intervention is based on the principles of the process of adaptation to retirement defined by Atchley and the Prochaska and Diclemente Model on the phases of preparation for retirement. The material to be used will be based on existing resources for retired people, awareness through multimedia material and knowledge of possible contributions of different technological devices to healthy-lifestyle.

ELIGIBILITY:
Inclusion criteria:

* People retired recently (since 10 years maximum)
* People who attend regularly the institution selected for recruitment, which is attended by retired people over the age of 60 years old.

Exclusion criteria:

* People who present cognitive and psychological alterations that may interfere in the interview
* People who have not had paid employment
* People who have completed previously a preparation for retirement's program.

Ages: 61 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in quality of life | Baseline and immediately after intervention (two months)
  EuroQol-5D: To measure the quality of life variable before and after intervention. This tool allows exploring the perception of each participant about their health status and quality of life. This scale measures three elements: A descriptive dimension divided into 5 dimensions: mobility, personal care, daily activities, pain/discomfort and anxiety/depression. The person must choose between one of the following levels of severity: 1 or absence of problems, 2 or presence of some problems, 3 or presence of serious or moderate problems. A visual analogue scale: the person indicates in a rule of 0 or worse health, to 100 or better health.

SECONDARY OUTCOMES:
Behavioural adopted in terms of retirement | One month before intervention
  It was measured according to the phase in which the person is at the beginning of the intervention, be it pre-contemplation in which the person is unaware of or uninterested in preparing and training for retirement, so he or she has no intention of changing his or her behavior; contemplation in which the person is aware of the possible difficulties he or she will have to face in the retirement stage, but does not assimilate the need to change his or her behavior; or action in which the person begins to think about different ideas for retirement and puts them into practice.
Changes in behavioural adopted in terms of retirement | Baseline and immediately after intervention (two months)
  It was measured according to the phase in which the person is at the end of the intervention, be it pre-contemplation in which the person is unaware of or uninterested in preparing and training for retirement, so he or she has no intention of changing his or her behavior; contemplation in which the person is aware of the possible difficulties he or she will have to face in the retirement stage, but does not assimilate the need to change his or her behavior; or action in which the person begins to think about different ideas for retirement and puts them into practice.
Individual-interviews | One month before intervention
  To know the individual experience about the stage before retirement, the moment of retirement, the present life, future expectations and the meaning of retirement.
Group-interviews | Immediately after intervention (1 month)
  To know the experience at group level of how they have lived the intervention, what it has brought them, how they have felt with the technology and what sense they give to it after carrying out the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Nieto-Riveiro, PhD, Principal Investigator — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan contains the collection of the variables extracted from the Euroqol-5D-5L scale and the sociodemographic data of the study sample, the study protocol developed, and the informed consent form used.

REFERENCES:
- [Background] Ye B, Chen H, Huang L, Ruan Y, Qi S, Guo Y, Huang Z, Sun S, Chen X, Shi Y, Gao J, Jiang Y. Changes in frailty among community-dwelling Chinese older adults and its predictors: evidence from a two-year longitudinal study. BMC Geriatr. 2020 Apr 10;20(1):130. doi: 10.1186/s12877-020-01530-x. PMID 32272903
- [Background] Gschwind YJ, Eichberg S, Ejupi A, de Rosario H, Kroll M, Marston HR, Drobics M, Annegarn J, Wieching R, Lord SR, Aal K, Vaziri D, Woodbury A, Fink D, Delbaere K. ICT-based system to predict and prevent falls (iStoppFalls): results from an international multicenter randomized controlled trial. Eur Rev Aging Phys Act. 2015 Nov 27;12:10. doi: 10.1186/s11556-015-0155-6. eCollection 2015. PMID 26865874
- [Background] Hamm JM, Heckhausen J, Shane J, Lachman ME. Risk of cognitive declines with retirement: Who declines and why? Psychol Aging. 2020 May;35(3):449-457. doi: 10.1037/pag0000453. Epub 2020 Mar 16. PMID 32175753
- [Background] Atchley RC. Adjustment to loss of job at retirement. Int J Aging Hum Dev. 1975;6(1):17-27. doi: 10.2190/EHU3-VCRV-VCRJ-04NU. PMID 1150332
- [Background] Atchley RC. The meaning of retirement. J Commun. 1974 Autumn;24(4):97-100. doi: 10.1111/j.1460-2466.1974.tb00414.x. No abstract available. PMID 4448858
- [Background] Park BH, Lee MS, Hong JY, Bae SH, Kim EY, Kim KK, Kim DK. The stages of physical activity and exercise behavior: an integrated approach to the theory of planned behavior. Asia Pac J Public Health. 2009 Jan;21(1):71-83. doi: 10.1177/1010539508327089. Epub 2008 Nov 17. PMID 19124338
- [Background] Pazzim TA, Marin AH. Retirement preparation program: evaluation of results. Psicol Reflex Crit. 2017 Dec 8;30(1):24. doi: 10.1186/s41155-017-0079-3. PMID 32026182
- [Background] Greig A, Dawes D, Murphy S, Parker G, Loveridge B. Program evaluation of a model to integrate internationally educated health professionals into clinical practice. BMC Med Educ. 2013 Oct 11;13:140. doi: 10.1186/1472-6920-13-140. PMID 24119470
- [Background] Ballesteros S, Kraft E, Santana S, Tziraki C. Maintaining older brain functionality: A targeted review. Neurosci Biobehav Rev. 2015 Aug;55:453-77. doi: 10.1016/j.neubiorev.2015.06.008. Epub 2015 Jun 6. PMID 26054789
- [Background] Hessel P. Does retirement (really) lead to worse health among European men and women across all educational levels? Soc Sci Med. 2016 Feb;151:19-26. doi: 10.1016/j.socscimed.2015.12.018. Epub 2015 Dec 15. PMID 26773290
- [Background] Brown RT, Diaz-Ramirez LG, Boscardin WJ, Lee SJ, Steinman MA. Functional Impairment and Decline in Middle Age: A Cohort Study. Ann Intern Med. 2017 Dec 5;167(11):761-768. doi: 10.7326/M17-0496. Epub 2017 Oct 31. PMID 29132150
- [Background] Klugar M, Cap J, Klugarova J, Mareckova J, Roberson DN, Kelnarova Z. The personal active aging strategies of older adults in Europe: a systematic review of qualitative evidence. JBI Database System Rev Implement Rep. 2016 May;14(5):193-257. doi: 10.11124/JBISRIR-2016-002393. PMID 27532471
- [Background] Damant J, Knapp M, Freddolino P, Lombard D. Effects of digital engagement on the quality of life of older people. Health Soc Care Community. 2017 Nov;25(6):1679-1703. doi: 10.1111/hsc.12335. Epub 2016 Feb 25. PMID 26919220
- See also: Official page of EuroQol Group who create the Quality of Life test. — https://euroqol.org/
- See also: Retired people association. — http://www.jubilares.es/
- See also: Data and analysis on population ageing. — http://www.globalagewatch.org/
- See also: Brief Intervention in Preparation for Retirement. — http://pepsic.bvsalud.org/scielo.php?script=sci_serial&pid=1679-3390&lng=pt&nrm=iso